CLINICAL TRIAL: NCT03930732
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, 52-week Pivotal Study to Assess the Efficacy, Safety and Tolerability of Dupilumab in Patients With Moderate-to-severe Chronic Obstructive Pulmonary Disease (COPD) With Type 2 Inflammation
Brief Title: Pivotal Study to Assess the Efficacy, Safety and Tolerability of Dupilumab in Patients With Moderate-to-severe COPD With Type 2 Inflammation
Acronym: BOREAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC15804; 2018-001953-28 (EudraCT Number); U1111-1211-8804 (Other: UTN)
Record Dates: First submitted 2019-04-26; First posted 2019-04-29 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dupilumab (Experimental): Participants received dupilumab 300 mg administered as SC injections q2w up to a maximum of 52 weeks (last dose administered at Week 50, EOT visit occurred 2 weeks after last administration of treatment i.e., at Week 52).
  Interventions: Drug: Dupilumab SAR231893; Drug: Inhaled Corticosteroid; Drug: Inhaled Long-Acting Beta Agonist; Drug: Inhaled Long-Acting Muscarinic Antagonist
- Placebo (Placebo Comparator): Participants received placebo matched to dupilumab 300 mg as subcutaneous (SC) injections q2w up to a maximum of 52 weeks (last dose administered at Week 50, end of treatment [EOT] visit occurred 2 weeks after last administration of treatment i.e., at Week 52).
  Interventions: Drug: Inhaled Corticosteroid; Drug: Inhaled Long-Acting Beta Agonist; Drug: Inhaled Long-Acting Muscarinic Antagonist; Drug: Placebo

INTERVENTIONS:
Drug: Dupilumab SAR231893 — Pharmaceutical form: Solution for injection
  Route of administration: Subcutaneous
  Other Names: Dupixent
  Arms: Dupilumab
Drug: Inhaled Corticosteroid — Pharmaceutical form: Inhaled Powder
  Route of administration: Oral inhalation
Drug: Inhaled Long-Acting Beta Agonist — Pharmaceutical form: Inhaled Powder
  Route of administration: Oral inhalation
Drug: Inhaled Long-Acting Muscarinic Antagonist — Pharmaceutical form: Inhaled Powder
  Route of administration: Oral inhalation
Drug: Placebo — Pharmaceutical form: Solution for injection
  Route of administration: Subcutaneous
  Arms: Placebo

SUMMARY:
Primary Objective:

To evaluate the efficacy of dupilumab administered every 2 weeks in patients with moderate-or severe Chronic Obstructive Pulmonary Disease (COPD) as measured by

* Annualized rate of acute moderate and severe COPD exacerbation (AECOPD)

Secondary Objectives:

To evaluate the effect of dupilumab administered every 2 weeks on

* Pre-bronchodilator forced expiratory volume in 1 second (FEV1) over 12 weeks compared to placebo
* Health related quality of life, assessed by the change from baseline to Week 52 in the St. George's Respiratory Questionnaire (SGRQ)
* Pre-bronchodilator FEV1 over 52 weeks compared to placebo
* Lung function assessments
* Moderate and severe COPD exacerbations
* To evaluate safety and tolerability
* To evaluate dupilumab systemic exposure and incidence of anti-drug antibodies (ADA)

DETAILED DESCRIPTION:
Approximately 68 weeks including a 4-week screening period, a 52-week treatment period, and 12 weeks of follow-up.

ELIGIBILITY:
Inclusion criteria:

* Participants with a physician diagnosis of COPD who met the following criteria at screening:

  * Current or former smokers with a smoking history of ≥10 pack-years.
  * Moderate-to-severe COPD (post-bronchodilator FEV1/ forced vital capacity [FVC] ratio <0.70 and post-bronchodilator FEV1 % predicted >30% and ≤70%).
  * Medical Research Council (MRC) Dyspnea Scale grade ≥2.
  * Patient-reported history of signs and symptoms of chronic bronchitis (chronic productive cough) for 3 months in the year up to screening in the absence of other known causes of chronic cough.
  * Documented history of high exacerbation risk defined as exacerbation history of ≥2 moderate or ≥1 severe within the year prior to inclusion. At least one exacerbation should have occurred while the patient was taking inhaled corticosteroid (ICS)/long acting beta agonist (LABA)/long acting muscarinic antagonist (LAMA) (or LABA/LAMA if ICS is contraindicated). Moderate exacerbations were recorded by the investigator and defined as acute exacerbation of COPD (AECOPD) that required either systemic corticosteroids (intramuscular, intravenous, or oral) and/or antibiotics. One of the two required moderate exacerbations had to require the use of systemic corticosteroids. Severe exacerbations were recorded by the investigator and defined as AECOPD requiring hospitalization or observation >24 hours in emergency department/urgent care facility.
  * Background triple therapy (ICS + LABA + LAMA) for 3 months prior to randomization with a stable dose of medication for ≥1 month prior to Visit 1; Double therapy (LABA + LAMA) allowed if ICS was contraindicated.
* Evidence of Type 2 inflammation: Patients with blood eosinophils ≥300 cells/microliter at Visit 1.

Exclusion criteria:

* COPD diagnosis for less than 12 months prior to randomization.
* A current diagnosis of asthma or history of asthma according to the 2018 Global Initiative for Asthma (GINA) guidelines or other accepted guidelines.
* Significant pulmonary disease other than COPD (e.g., lung fibrosis, sarcoidosis, interstitial lung disease, pulmonary hypertension, bronchiectasis, Churg-Strauss Syndrome etc) or another diagnosed pulmonary or systemic disease associated with elevated peripheral eosinophil counts.
* Cor pulmonale, evidence of right cardiac failure.
* Treatment with oxygen of more than 12 hours per day.
* Hypercapnia requiring Bi-level ventilation.
* AECOPD as defined in inclusion criteria within 4 weeks prior to screening, or during the screening period.
* Respiratory tract infection within 4 weeks prior to screening, or during the screening period.
* History of, or planned pneumonectomy or lung volume reduction surgery. Patients who were participating in the acute phase of a pulmonary rehabilitation program, ie, who started rehabilitation <4 weeks prior to screening (Note: patients in the maintenance phase of a rehabilitation program could be included).
* Diagnosis of α-1 anti-trypsin deficiency.

The above information was not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 939 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (275):
- United States (51):
  - SEC Clinical Research, LLC-Site Number:8400030, Andalusia, Alabama
  - Clinical Research Center of Alabama, LLC-Site Number:8400041, Birmingham, Alabama
  - UAB Lung Health Center-Site Number:8400013, Birmingham, Alabama
  - SEC Clinical Research, LLC-Site Number:8400059, Dothan, Alabama
  - Pulmonary Associates of Mobile, P.C.-Site Number:8400057, Mobile, Alabama
  - Asthma and Allergy Associates, PC-Site Number:8400034, Colorado Springs, Colorado
  - Clinical Research Of West Florida Inc-Site Number:8400010, Clearwater, Florida
  - Finlay Medical Research-Site Number:8400014, Greenacres City, Florida
  - Project 4 research, Inc.-Site Number:8400023, Miami, Florida
  - Finlay Medical Research-Site Number:8400062, Miami, Florida
  - Renstar Medical Research-Site Number:8400051, Ocala, Florida
  - Florida Institute for Clinical Research, LLC-Site Number:8400029, Orlando, Florida
  - Emerald Coast Research Associates-Site Number:8400032, Panama City, Florida
  - Sarasota Clinical Research-Site Number:8400026, Sarasota, Florida
  - VitaLink research-Hamilton Mill-Site Number:8400055, Dacula, Georgia
  - DC Research Works-Site Number:8400016, Marietta, Georgia
  - North Georgia Clinical Research-Site Number:8400025, Woodstock, Georgia
  - Johns Hopkins University (Asthma and Allergy Center)-Site Number:8400012, Baltimore, Maryland
  - Asthma Allergy & Sinus Center-Site Number:8400038, White Marsh, Maryland
  - Michigan Medicine (University of Michigan)-Site Number:8400050, Ann Arbor, Michigan
  - Mayo Clinic Lanmark Center 2-46-Site Number:8400065, Rochester, Minnesota
  - Midwest Chest Consultants, P.C.-Site Number:8400011, Saint Charles, Missouri
  - Washington University School of Medicine-Site Number:8400004, St Louis, Missouri
  - Sierra Clinical Research-Site Number:8400035, Las Vegas, Nevada
  - Va Western New York Healthcare-Site Number:8400067, Buffalo, New York
  - IMA Clinical Research, LLC-Site Number:8400070, New York, New York
  - The University of North Carolina at Chapel Hill - Division of Pulmonary and Critical Care Medicine-Site Number:8400019, Chapel Hill, North Carolina
  - American Health Research-Site Number:8400061, Charlotte, North Carolina
  - Duke Asthma, Allergy and Airway Center-Site Number:8400064, Durham, North Carolina
  - Accellacare-Site Number:8400052, Wilmington, North Carolina
  - Southeastern Research Center-Site Number:8400060, Winston-Salem, North Carolina
  - Midwest Pulmonary and Sleep Research Center-Site Number:8400040, Dayton, Ohio
  - Aventiv Research, Inc-Site Number:8400024, Dublin, Ohio
  - OK Clinical Research-Site Number:8400005, Edmond, Oklahoma
  - Velocity Clinical Research, Medford-Site Number:8400001, Medford, Oregon
  - Jefferson Associates in Internal Medicine-Site Number:8400037, Clairton, Pennsylvania
  - Temple University Hospital-Site Number:8400009, Philadelphia, Pennsylvania
  - Emphysema COPD Research Center, Kaufmann Medical Building-Site Number:8400033, Pittsburgh, Pennsylvania
  - Berks Schuylkill Respiratory Specialists, LTD-Site Number:8400063, Wyomissing, Pennsylvania
  - VitaLink Research-Easley-Site Number:8400022, Easley, South Carolina
  - VitaLink Research- Gaffney-Site Number:8400047, Gaffney, South Carolina
  - VitaLink Research-Greenville-Site Number:8400007, Greenville, South Carolina
  - Clinical Research of Charleston-Site Number:8400044, Mt. Pleasant, South Carolina
  - Clinical Research of Rock Hill-Site Number:8400046, Rock Hill, South Carolina
  - VitaLink Research - Spartanburg-Site Number:8400048, Spartanburg, South Carolina
  - Clinical Trials Center of Middle Tennessee-Site Number:8400073, Franklin, Tennessee
  - Bayer College of Medicine-Site Number:8400018, Houston, Texas
  - Metroplex Pulmonary and Sleep Center-Site Number:8400021, McKinney, Texas
  - Sherman Clinical Research-Site Number:8400027, Sherman, Texas
  - MultiCare Institute for Research and Innovation-Site Number:8400036, Tacoma, Washington
  - Allergy, Asthma & Sinus Center, S.C.-Site Number:8400008, Greenfield, Wisconsin
- Argentina (12):
  - Investigational Site Number :0320011, CABA, Buenos Aires
  - Investigational Site Number :0320002, CABA, Buenos Aires
  - Investigational Site Number :0320003, CABA, Buenos Aires
  - Investigational Site Number :0320004, CABA, Buenos Aires
  - Investigational Site Number :0320012, La Plata, Buenos Aires
  - Investigational Site Number :0320007, Quilmes, Buenos Aires F.D.
  - Investigational Site Number :0320006, Rosario, Santa Fe Province
  - Investigational Site Number :0320009, San Miguel de Tucumán, Tucumán Province
  - Investigational Site Number :0320001, Buenos Aires
  - Investigational Site Number :0320005, Buenos Aires
  - Investigational Site Number :0320008, Mar del Plata
  - Investigational Site Number :0320010, Mendoza
- Bulgaria (8):
  - Investigational Site Number :1001004, Haskovo
  - Investigational Site Number :1001003, Montana
  - Investigational Site Number :1001006, Rousse
  - Investigational Site Number :1001009, Sofia
  - Investigational Site Number :1001002, Sofia
  - Investigational Site Number :1001001, Sofia
  - Investigational Site Number :1001005, Stara Zagora
  - Investigational Site Number :1001010, Troyan Municipality
- Canada (20):
  - Investigational Site Number :1240021, Edmonton, Alberta
  - Investigational Site Number :1240015, Edmonton, Alberta
  - Investigational Site Number :1240016, Sherwood Park, Alberta
  - Investigational Site Number :1240017, Vancouver, British Columbia
  - Investigational Site Number :1240007, Vancouver, British Columbia
  - Investigational Site Number :1240002, Burlington, Ontario
  - Investigational Site Number :1240012, Toronto, Ontario
  - Investigational Site Number :1240013, Windsor, Ontario
  - Investigational Site Number :1240009, Montreal, Quebec
  - Investigational Site Number :1240003, Montreal, Quebec
  - Investigational Site Number :1240001, Montreal, Quebec
  - Investigational Site Number :1240010, Sherbrooke, Quebec
  - Investigational Site Number :1240011, Sherbrooke, Quebec
  - Investigational Site Number :1240006, St-charles Borrommee, Quebec
  - Investigational Site Number :1240008, Trois-Rivières, Quebec
  - Investigational Site Number :1240020, Victoriaville, Quebec
  - Investigational Site Number :1240005, Québec
  - Investigational Site Number :1240004, Québec
  - Investigational Site Number :1240019, Québec
  - Investigational Site Number :1240018, Québec
- Chile (8):
  - Investigational Site Number :1520006, Curicó, Maule Region
  - Investigational Site Number :1520001, Talca, Maule Region
  - Investigational Site Number :1520009, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number :1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number :1520005, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number :1520008, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number :1520002, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number :1520004, Quillota, Región de Valparaíso
- China (37):
  - Investigational Site Number :1560037, Baotou
  - Investigational Site Number :1560006, Beijing
  - Investigational Site Number :1560003, Changchun
  - Investigational Site Number :1560022, Changsha
  - Investigational Site Number :1560021, Changsha
  - Investigational Site Number :1560001, Chengdu
  - Investigational Site Number :1560017, Chengdu
  - Investigational Site Number :1560012, Chongqing
  - Investigational Site Number :1560005, Chongqing
  - Investigational Site Number :1560053, Fuzhou
  - Investigational Site Number :1560036, Guangzhou
  - Investigational Site Number :1560019, Guangzhou
  - Investigational Site Number :1560045, Haikou
  - Investigational Site Number :1560018, Haikou
  - Investigational Site Number :1560046, Hangzhou
  - Investigational Site Number :1560009, Hefei
  - Investigational Site Number :1560041, Hefei
  - Investigational Site Number :1560015, Hohhot
  - Investigational Site Number :1560008, Hohhot
  - Investigational Site Number :1560027, Nanchang
  - Investigational Site Number :1560034, Nanjing
  - Investigational Site Number :1560032, Shanghai
  - Investigational Site Number :1560013, Shanghai
  - Investigational Site Number :1560007, Shanghai
  - Investigational Site Number :1560014, Shenyang
  - Investigational Site Number :1560004, Shenyang
  - Investigational Site Number :1560051, Shenzhen
  - Investigational Site Number :1560016, Shijiazhuang
  - Investigational Site Number :1560024, Taiyuan
  - Investigational Site Number :1560010, Tianjin
  - Investigational Site Number :1560028, Ürümqi
  - Investigational Site Number :1560052, Wuhan
  - Investigational Site Number :1560020, Xi'an
  - Investigational Site Number :1560054, Xuzhou
  - Investigational Site Number :1560011, Yangzhou
  - Investigational Site Number :1560031, Zhanjiang
  - Investigational Site Number :1560002, Zhengzhou
- Czechia (8):
  - Investigational Site Number :2030002, Jindrichuv Hradec III
  - Investigational Site Number :2030005, Karlovy Vary
  - Investigational Site Number :2030009, Miroslav
  - Investigational Site Number :2030001, Nový Bor
  - Investigational Site Number :2030003, Prague
  - Investigational Site Number :2030008, Praha 6 - Brevnov
  - Investigational Site Number :2030004, Rokycany
  - Investigational Site Number :2030006, Strakonice
- Denmark (7):
  - Investigational Site Number :2080003, Aalborg
  - Investigational Site Number :2080001, Copenhagen Nv
  - Investigational Site Number :2080002, Hvidovre
  - Investigational Site Number :2080006, Næstved
  - Investigational Site Number :2080005, Odense C
  - Investigational Site Number :2080004, Roskilde
  - Investigational Site Number :2080007, Vejle
- Finland (2):
  - Investigational Site Number :2460003, Pori
  - Investigational Site Number :2460001, Turku
- Germany (7):
  - Investigational Site Number :2760006, Berlin
  - Investigational Site Number :2760009, Frankfurt am Main
  - Investigational Site Number :2760002, Hamburg
  - Investigational Site Number :2760007, Koblenz
  - Investigational Site Number :2760011, Leipzig
  - Investigational Site Number :2760010, Lübeck
  - Investigational Site Number :2760008, Marburg
- Hungary (11):
  - Investigational Site Number :3480007, Balassagyarmat
  - Investigational Site Number :3480011, Budapest
  - Investigational Site Number :3480008, Edelény
  - Investigational Site Number :3480001, Gödöllö
  - Investigational Site Number :3480010, Hajdunánás
  - Investigational Site Number :3480002, Komárom
  - Investigational Site Number :3480003, Makó
  - Investigational Site Number :3480006, Mohács
  - Investigational Site Number :3480012, Püspökladány
  - Investigational Site Number :3480004, Százhalombatta
  - Investigational Site Number :3480005, Szombathely
- Israel (7):
  - Investigational Site Number :3760006, Ashkelon
  - Investigational Site Number :3760007, Beersheba
  - Investigational Site Number :3760003, Haifa
  - Investigational Site Number :3760005, Jerusalem
  - Investigational Site Number :3760004, Jerusalem
  - Investigational Site Number :3760001, Petah Tikva
  - Investigational Site Number :3760002, Rehovot
- Italy (5):
  - Investigational Site Number :3800004, Cona, Ferrara
  - Investigational Site Number :3800003, Rozzano, Milano
  - Investigational Site Number :3800007, Pisa
  - Investigational Site Number :3800001, Reggio Emilia
  - Investigational Site Number :3800005, Roma
- Japan (22):
  - Investigational Site Number :3920013, Kasuga-shi, Fukuoka
  - Investigational Site Number :3920011, Himeji-shi, Hyōgo
  - Investigational Site Number :3920023, Higashiibaraki-gun, Ibaraki
  - Investigational Site Number :3920014, Naka-gun, Ibaraki
  - Investigational Site Number :3920019, Takamatsu, Kagawa-ken
  - Investigational Site Number :3920027, Yokohama, Kanagawa
  - Investigational Site Number :3920003, Joyo-shi, Kyoto
  - Investigational Site Number :3920017, Kyoto, Kyoto
  - Investigational Site Number :3920006, Ueda-shi, Nagano
  - Investigational Site Number :3920029, Urasoe-shi, Okinawa
  - Investigational Site Number :3920018, Kawachinagano-shi, Osaka
  - Investigational Site Number :3920001, Kishiwada-shi, Osaka
  - Investigational Site Number :3920028, Osaka, Osaka
  - Investigational Site Number :3920012, Sakai-shi, Osaka
  - Investigational Site Number :3920021, Hamamatsu, Shizuoka
  - Investigational Site Number :3920008, Chuo-ku, Tokyo
  - Investigational Site Number :3920030, Chuo-ku, Tokyo
  - Investigational Site Number :3920005, Chuo-ku, Tokyo
  - Investigational Site Number :3920015, Kokubunji-shi, Tokyo
  - Investigational Site Number :3920016, Shinagawa-ku, Tokyo
  - Investigational Site Number :3920004, Toshima-ku, Tokyo
  - Investigational Site Number :3920026, Toshima-ku, Tokyo
- Mexico (7):
  - Investigational Site Number :4840002, Guadalajara, Jalisco
  - Investigational Site Number :4840001, Monterrey, Nuevo León
  - Investigational Site Number :4840004, Chihuahua City
  - Investigational Site Number :4840003, Durango
  - Investigational Site Number :4840006, Mexico City
  - Investigational Site Number :4840007, Oaxaca City
  - Investigational Site Number :4840005, Veracruz
- Poland (9):
  - Investigational Site Number :6160016, Poznan, Greater Poland Voivodeship
  - Investigational Site Number :6160006, Poznan, Greater Poland Voivodeship
  - Investigational Site Number :6160009, Grudziądz, Kuyavian-Pomeranian Voivodeship
  - Investigational Site Number :6160007, Krakow, Lesser Poland Voivodeship
  - Investigational Site Number :6160015, Grodzisk Mazowiecki, Masovian Voivodeship
  - Investigational Site Number :6160012, Warsaw, Masovian Voivodeship
  - Investigational Site Number :6160008, Bialystok, Podlaskie Voivodeship
  - Investigational Site Number :6160014, Elblag, Pomeranian Voivodeship
  - Investigational Site Number :6160011, Katowice, Silesian Voivodeship
- Romania (8):
  - Investigational Site Number :6420001, Bucharest
  - Investigational Site Number :6420009, Bucharest
  - Investigational Site Number :6420008, Bucharest
  - Investigational Site Number :6420003, Cluj-Napoca
  - Investigational Site Number :6420004, Cluj-Napoca
  - Investigational Site Number :6420007, Constanța
  - Investigational Site Number :6420006, Timișoara
  - Investigational Site Number :6420010, Timișoara
- Russia (9):
  - Investigational Site Number :6430003, Chelyabinsk
  - Investigational Site Number :6430004, Kazan'
  - Investigational Site Number :6430006, Moscow
  - Investigational Site Number :6430001, Moscow
  - Investigational Site Number :6430005, Moscow
  - Investigational Site Number :6430008, Moscow
  - Investigational Site Number :6430002, Moscow
  - Investigational Site Number :6430009, Moscow
  - Investigational Site Number :6430007, Saint Petersburg
- Slovakia (5):
  - Investigational Site Number :7030007, Banská Bystrica
  - Investigational Site Number :7030006, Humenné
  - Investigational Site Number :7030003, Levice
  - Investigational Site Number :7030001, Poprad
  - Investigational Site Number :7030002, Spišská Nová Ves
- South Korea (6):
  - Investigational Site Number :4100003, Wŏnju, Gangwon-do
  - Investigational Site Number :4100004, Seongnam-si, Gyeonggi-do
  - Investigational Site Number :4100008, Incheon, Incheon-gwangyeoksi
  - Investigational Site Number :4100001, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number :4100009, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number :4100007, Seoul, Seoul-teukbyeolsi
- Spain (9):
  - Investigational Site Number :7240096, Santiago de Compostela, A Coruña [La Coruña]
  - Investigational Site Number :7240002, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number :7240007, Sant Boi de Llobregat, Barcelona [Barcelona]
  - Investigational Site Number :7240005, Mérida / Badajoz, Extremadura
  - Investigational Site Number :7240006, Pozuelo de Alarcón, Madrid
  - Investigational Site Number :7240003, Madrid
  - Investigational Site Number :7240001, Málaga
  - Investigational Site Number :7240010, Palma de Mallorca
  - Investigational Site Number :7240004, Valencia
- Sweden (2):
  - Investigational Site Number :7520001, Lund
  - Investigational Site Number :7520002, Stockholm
- Turkey (Türkiye) (7):
  - Investigational Site Number :7920004, Ankara
  - Investigational Site Number :7920001, Istanbul
  - Investigational Site Number :7920006, Izmir
  - Investigational Site Number :7920007, Izmir
  - Investigational Site Number :7920008, Kırıkkale
  - Investigational Site Number :7920005, Manisa
  - Investigational Site Number :7920002, Mersin
- Ukraine (8):
  - Investigational Site Number :8040003, Chernivtsi
  - Investigational Site Number :8040001, Ivano-Frankivsk
  - Investigational Site Number :8040006, Kharkiv
  - Investigational Site Number :8040004, Kyiv
  - Investigational Site Number :8040009, Odesa
  - Investigational Site Number :8040002, Ternopil
  - Investigational Site Number :8040005, Vinnytsia
  - Investigational Site Number :8040007, Zhytomyr

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Christenson SA, Hanania NA, Bhatt SP, Bafadhel M, Rabe KF, Vogelmeier CF, Papi A, Singh D, Laws E, Dakin P, Bansal A, Lu X, Bauer D, Maloney J, Robinson LB, Abdulai RM. Type 2 inflammation biomarkers and their association with response to dupilumab in COPD (BOREAS): an analysis of a randomised, placebo-controlled, phase 3 trial. Lancet Respir Med. 2025 Aug;13(8):687-697. doi: 10.1016/S2213-2600(25)00044-X. Epub 2025 Jul 9. PMID 40651490
- [Derived] Vogelmeier CF, Rabe KF, Bhatt SP, Hanania NA, Bafadhel M, Christenson SA, Papi A, Singh D, Laws E, Maloney J, Dakin P, Lu X, Bauer D, Bansal A, Robinson LB, Abdulai RM. Dupilumab reduces acute exacerbations and improves lung function in patients with COPD with type 2 inflammation irrespective of body mass index, airflow obstruction, dyspnea, and exercise capacity index scores. Respir Med. 2025 May;241:108015. doi: 10.1016/j.rmed.2025.108015. Epub 2025 Feb 28. PMID 40024335
- [Derived] Bhatt SP, Rabe KF, Hanania NA, Vogelmeier CF, Bafadhel M, Christenson SA, Papi A, Singh D, Laws E, Dakin P, Maloney J, Lu X, Bauer D, Bansal A, Abdulai RM, Robinson LB. Effect of Dupilumab on Health-Related Quality of Life and Respiratory Symptoms in Patients With COPD and Type 2 Inflammation: BOREAS and NOTUS. Chest. 2025 Jul;168(1):56-66. doi: 10.1016/j.chest.2025.01.029. Epub 2025 Jan 31. PMID 39894389
- [Derived] Bhatt SP, Rabe KF, Hanania NA, Vogelmeier CF, Bafadhel M, Christenson SA, Papi A, Singh D, Laws E, Dakin P, Maloney J, Lu X, Bauer D, Bansal A, Robinson LB, Abdulai RM. Dupilumab reduces exacerbations and improves lung function in patients with chronic obstructive pulmonary disease and emphysema: Phase 3 randomized trial (BOREAS). Respir Med. 2025 Jan;236:107846. doi: 10.1016/j.rmed.2024.107846. Epub 2024 Oct 30. PMID 39481660
- [Derived] Bhatt SP, Rabe KF, Hanania NA, Vogelmeier CF, Cole J, Bafadhel M, Christenson SA, Papi A, Singh D, Laws E, Mannent LP, Patel N, Staudinger HW, Yancopoulos GD, Mortensen ER, Akinlade B, Maloney J, Lu X, Bauer D, Bansal A, Robinson LB, Abdulai RM; BOREAS Investigators. Dupilumab for COPD with Type 2 Inflammation Indicated by Eosinophil Counts. N Engl J Med. 2023 Jul 20;389(3):205-214. doi: 10.1056/NEJMoa2303951. Epub 2023 May 21. PMID 37272521

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 275 centers in 24 countries. A total of 2599 participants were screened from 15 Apr 2019 to 12 Jan 2022, of which 1660 were screen failures due to not meeting eligibility criteria.
Pre-assignment Details: A total of 939 participants were randomized in a 1:1 ratio to receive either dupilumab 300 milligrams (mg) every 2 weeks (q2w) or matching placebo for 52 weeks.
Groups:
- Dupilumab 300 mg q2w: Participants received dupilumab 300 mg administered as SC injections q2w up to a maximum of 52 weeks (last dose administered at Week 50, EOT visit occurred 2 weeks after last administration of treatment i.e., at Week 52).
Period: Overall Study
Arm/Group | Placebo | Dupilumab 300 mg q2w
Started (Randomized) | 471 | 468
Safety Population (One participant was exposed to different treatment other than planned (was randomized to placebo arm but received dupilumab on Day 40). The actual arm was considered as dupilumab 300 mg q2w. In safety analyses, the actual arms are used.) | 470 | 469
Completed | 434 | 440
Not Completed | 37 | 28
Not completed — Adverse Event | 9 | 7
Not completed — Poor compliance to protocol | 0 | 1
Not completed — Withdrawal by Subject | 23 | 11
Not completed — Other reason related to Coronavirus Disease-2019 (COVID-19) | 0 | 1
Not completed — Other reason not related to COVID-19 | 5 | 8

BASELINE CHARACTERISTICS:
Population: The Randomized population consisted of any participant who was allocated to a randomized treatment regardless of whether the treatment kit was used.
Groups:
- Placebo: Participants received placebo matched to dupilumab 300 mg as SC injections q2w up to a maximum of 52 weeks (last dose administered at Week 50, EOT visit occurred 2 weeks after last administration of treatment i.e., at Week 52).
- Total: Total of all reporting groups
Arm/Group | Placebo | Dupilumab 300 mg q2w | Total
Number analyzed (Participants) | 471 | 468 | 939
Age, Continuous [Median (Standard Deviation); unit: years] | 65.2 (8.1) | 65.0 (8.0) | 65.1 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 170 | 319
  Male | 322 | 298 | 620
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 3 | 7
  Asian | 67 | 67 | 134
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 3 | 5
  White | 397 | 393 | 790
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Annualized Rate of Moderate or Severe Chronic Obstructive Pulmonary Disease (COPD) Exacerbations Over the 52-Week Treatment Period
Description: Moderate exacerbations were recorded by the Investigator and defined as acute exacerbation of COPD (AECOPD) that required either systemic corticosteroids (such as intramuscular, intravenous or oral) and/or antibiotics. Severe exacerbations were also recorded by the Investigator and defined as AECOPD requiring hospitalization, or observation for >24 hours in an emergency department/urgent care facility or resulting in death. For both moderate and severe events to be counted as separate events, they were separated by at least 14 days. Annualized event rate was the total number of exacerbations that occurred during the treatment period divided by the total number of participant-years treated. Events were adjudicated by independent third party.
Time Frame: Baseline (Day 1) to Week 52
Population: The intent-to-treat (ITT) population consisted of the randomized population analyzed according to the treatment group allocated by randomization.
Measure: Number (95% Confidence Interval); unit: exacerbation per participant-year
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 471 | 468
exacerbation per participant-year | 1.01 [0.931 to 1.301] | 0.776 [0.645 to 0.934]
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; Derived using negative binomial model with the total number of the events occurring during the 52-week treatment period as the response variable, and treatment group, region (pooled country), inhaled corticosteroid (ICS) dose, smoking status at screening, baseline disease severity, and number of moderate or severe COPD exacerbation events within one year prior to the study as covariates, and log-transformed treatment duration as an offset variable; Test type: Superiority — A hierarchical testing procedure was used to control type I error and handle primary and a few secondary endpoint analyses at a 2-sided significance level of 0.049. Testing was then performed sequentially in the order the endpoints are reported (till OM 9). The hierarchical testing sequence continued only when the previous endpoint was statistically significant at 0.049 level; p = 0.0005, Negative binomial model; Risk Difference (RD) = -0.324, 95% CI 2-sided [-0.508 to -0.140] — Derived using delta method

2. Secondary Outcome: Change From Baseline in Pre-Bronchodilator (BD) Forced Expiratory Volume in One Second (FEV1) at Week 12
Description: The FEV1 was the volume of air exhaled from the lungs in the first second of a forced expiration as measured by spirometer. Spirometry was performed after a wash out period of bronchodilators according to their action duration.
Time Frame: Baseline (Day 1) to Week 12
Population: The ITT population consisted of the randomized population analyzed according to the treatment group allocated by randomization. Only those participants with data available were analyzed.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 469 | 466
liters | 0.077 (0.018) | 0.160 (0.018)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; Derived from mixed-effect model with repeated measures (MMRM) model with the change from baseline in pre-BD FEV1 up to Week 12 as response variables, and treatment group, age, sex, height, region (pooled country), ICS dose, smoking status at screening, visit, treatment-by-visit interaction, baseline pre-BD FEV1, and FEV1 baseline-by-visit interaction as covariates. Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant); Test type: Superiority; p < 0.0001, MMRM model — Threshold for significance at 0.049 level; Least Square (LS) Mean Difference = 0.083, 95% CI 2-sided [0.042 to 0.125]

3. Secondary Outcome: Change From Baseline in Pre-BD FEV1 at Week 52
Description: as for outcome 2
Time Frame: Baseline (Day 1) to Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 469 | 466
liters | 0.070 (0.019) | 0.153 (0.019)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; Derived from MMRM model with the change from baseline in pre-BDFEV1 up to Week 52 as response variables, and treatment group, age, sex, height, region (pooled country), ICS dose, smoking status at screening, visit, treatment-by-visit interaction, baseline pre-BD FEV1, and FEV1 baseline-by-visit interaction as covariates. Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant); Test type: Superiority; p = 0.0003, MMRM model — Threshold for significance at 0.049 level; LS Mean Difference = 0.083, 95% CI 2-sided [0.038 to 0.128]

4. Secondary Outcome: Change From Baseline in Pre-BD FEV1 at Week 12 in Subgroup of Participants With Baseline Fractional Exhaled Nitric Oxide (FeNO) >=20 Parts Per Billion (Ppb)
Description: FeNO is a demonstrated biomarker of type 2 airway inflammation in respiratory diseases. FeNO was analyzed using a NIOX instrument or similar analyzer using a flow rate of 50 milliliter per second (mL/s) and reported in ppb. This assessment was conducted prior to spirometry and following a fast of at least 1 hour.
Time Frame: Baseline (Day 1) to Week 12
Population: The subgroup of participants with baseline FeNO >=20 ppb within the ITT population were included. Only those participants with data available were analyzed.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 186 | 193
liters | 0.108 (0.035) | 0.232 (0.034)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; Derived from MMRM model with the change from baseline in pre-BD FEV1 up to Week 12 as response variables, and treatment group, age, sex, height, region (pooled country), ICS dose, smoking status at screening, visit, treatment-by-visit interaction, baseline pre-BD FEV1, and FEV1 baseline-by-visit interaction as covariates. Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant); Test type: Superiority; p = 0.0022, MMRM model — Threshold for significance at 0.049 level; LS Mean Difference = 0.124, 95% CI 2-sided [0.045 to 0.203]

5. Secondary Outcome: Change From Baseline in Pre-BD FEV1 at Week 52 in Subgroup of Participants With Baseline FeNO >=20 Ppb
Description: FeNO is a demonstrated biomarker of type 2 airway inflammation in respiratory diseases. FeNO was analyzed using a NIOX instrument or similar analyzer using a flow rate of 50 mL/s and reported in ppb. This assessment was conducted prior to spirometry and following a fast of at least 1 hour.
Time Frame: Baseline (Day 1) to Week 52
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 186 | 193
liters | 0.120 (0.037) | 0.247 (0.036)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; Derived from MMRM model with the change from baseline in pre-BD FEV1 up to Week 52 as response variables, and treatment group, age, sex, height, region (pooled country), ICS dose, smoking status at screening, visit, treatment-by-visit interaction, baseline pre-BD FEV1, and FEV1 baseline-by-visit interaction as covariates. Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant); Test type: Superiority; p = 0.0034, MMRM model — Threshold for significance at 0.049 level; LS Mean Difference = 0.127, 95% CI 2-sided [0.042 to 0.212]

6. Secondary Outcome: Change From Baseline in Saint (St.) George's Respiratory Questionnaire (SGRQ) Total Score at Week 52
Description: The SGRQ was a 50-item self-administered questionnaire designed to measure and quantify health status in adult participants with chronic airflow limitation and rated on electronic diary. Scores by dimension were calculated for 3 domains: symptoms, activity and impacts (psycho-social) as well as a total score. Global and domain scores range from 0 to 100, with 100 representing the worst possible health status and 0 indicating the best possible health status. Higher score indicates worse health status/heath related quality of life.
Time Frame: Baseline (Day 1) to Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 456 | 456
score on a scale | -6.369 (0.816) | -9.732 (0.810)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; Derived from MMRM model with the change from baseline in SGRQ total score up to Week 52 as response variables, and treatment group, region (pooled country), ICS dose, smoking status at screening, treatment-by-visit interaction, baseline SGRQ total score, and SGRQ baseline-by-visit interaction as covariates. Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant); Test type: Superiority; p = 0.0017, MMRM model — Threshold for significance at 0.049 level; LS Mean Difference = -3.363, 95% CI 2-sided [-5.459 to -1.266]

7. Secondary Outcome: Percentage of Participants With SGRQ Improvement >=4 Points at Week 52
Description: A responder was defined as a participant with improvement from baseline in SGRQ total score at Week 52 by >=4 points. Participants with improvement <4 points or with missing values were considered as non-responders. The percentage of participants who achieved a clinically meaningful response in SGRQ total score (reduction [improvement] by >=4 points)/responders are reported.
Time Frame: Baseline (Day 1) to Week 52
Population: The ITT population consisted of the randomized population analyzed according to the treatment group allocated by randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 471 | 468
percentage of participants | 43.1 | 51.5
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; Derived from logistic regression model which includes treatment group, region (pooled country), ICS dose, smoking status at screening, and baseline SGRQ total score as covariates. Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant); Test type: Superiority; p = 0.0089, Regression, Logistic — Threshold for significance at 0.049 level; Odds Ratio (OR) = 1.439, 95% CI 2-sided [1.096 to 1.890]

8. Secondary Outcome: Change From Baseline in Evaluating Respiratory Symptoms (E-RS) in COPD (E-RS: COPD) RS-Total Score at Week 52
Description: The E-RS in COPD scale was a part of the exacerbations of chronic pulmonary disease tool (EXACT). It was a derivative instrument used to measure the effect of treatment on the severity of respiratory symptoms in stable COPD. E-RS: COPD RS-Total Score was derived based on weekly averages of daily assessed 11 respiratory symptom items contained in the 14-item EXACT questionnaire. The RS-Total score represented overall respiratory symptom severity, ranged from 0 to 40. Summation procedure was used to derive the three daily domain scores: 1). RS-Breathlessness (range 0-17), 2) RS-Cough and Sputum (score range 0-11), 3) RS-Chest Symptoms (score range 0-12). The higher the score, more severe were the symptoms.
Time Frame: Baseline (Day 1) to Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 467 | 461
score on a scale | -1.558 (0.256) | -2.694 (0.257)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; Derived from MMRM model with the change from baseline in E-RS: COPD RS-Total Score to Week 52 as response variables, and treatment group, region (pooled country), ICS dose, smoking status at screening, visit, treatment-by-visit interaction, baseline E-RS: COPD RS-Total Score, and baseline E-RS: COPD RS-Total Score-by-visit interaction as covariates. Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant); Test type: Superiority; p = 0.0012, MMRM model — Threshold for significance at 0.049 level; LS Mean Difference = -1.137, 95% CI 2-sided [-1.823 to -0.450]

9. Secondary Outcome: Annualized Rate of Moderate or Severe COPD Exacerbation Over the 52-Week Treatment Period in Subgroup of Participants With Baseline FeNO >=20 Ppb
Description: Moderate exacerbations were recorded by the Investigator and defined as AECOPD that required either systemic corticosteroids (such as intramuscular, intravenous or oral) and/or antibiotics. Severe exacerbations were also recorded by the investigator and defined as AECOPD requiring hospitalization, or observation for >24 hours in an emergency department/urgent care facility or resulting in death. For both moderate and severe events to be counted as separate events, they were separated by at least 14 days. Annualized event rate among participants with baseline FeNO >=20 ppb was the total number of exacerbations that occurred during the treatment period divided by the total number of participant-years treated. Events were adjudicated by independent third party.
Time Frame: Baseline (Day 1) to Week 52
Population: The subgroup of participants with baseline FeNO >=20 ppb within the ITT population were included.
Measure: Number (95% Confidence Interval); unit: exacerbation per participant-year
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 188 | 195
exacerbation per participant-year | 1.117 [0.831 to 1.502] | 0.699 [0.510 to 0.958]
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; Derived using negative binomial model with the total number of the events occurring during the 52-week treatment period as the response variable, and treatment group, region (pooled country), ICS dose, smoking status at screening, baseline disease severity, and number of moderate or severe COPD exacerbation events within one year prior to the study as covariates, and log-transformed treatment duration as an offset variable; Test type: Superiority — Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant); p = 0.0052, Negative binomial model — Threshold for significance at 0.049 level; Risk Difference (RD) = -0.418, 95% CI 2-sided [-0.728 to -0.109] — Derived using delta method

10. Secondary Outcome: Change From Baseline in Pre-BD FEV1 to Weeks 2, 4, 8, 24, 36 and 44
Description: as for outcome 2
Time Frame: Baseline (Day 1) to Weeks 2, 4, 8, 24, 36 and 44
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 469 | 466
liters
  Week 2 | 0.075 (0.017) | 0.159 (0.017)
  Week 4 | 0.069 (0.017) | 0.163 (0.017)
  Week 8 | 0.069 (0.017) | 0.149 (0.017)
  Week 24 | 0.068 (0.018) | 0.170 (0.018)
  Week 36 | 0.072 (0.018) | 0.155 (0.018)
  Week 44 | 0.089 (0.019) | 0.176 (0.019)

11. Secondary Outcome: Change From Baseline in Post-BD FEV1 to Weeks 2, 4, 8, 12, 24, 36 and 52
Description: The FEV1 was the volume of air exhaled from the lungs in the first second of a forced expiration as measured by spirometer. Post-BD FEV1 referred to the spirometry performed within 30 minutes after administration of bronchodilator.
Time Frame: Baseline (Day 1) to Weeks 2, 4, 8, 12, 24, 36 and 52
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 469 | 467
liters
  Week 2 | 0.071 (0.017) | 0.158 (0.017)
  Week 4 | 0.080 (0.017) | 0.158 (0.017)
  Week 8 | 0.077 (0.018) | 0.153 (0.018)
  Week 12 | 0.084 (0.018) | 0.156 (0.018)
  Week 24 | 0.072 (0.019) | 0.169 (0.019)
  Week 36 | 0.072 (0.019) | 0.155 (0.019)
  Week 52 | 0.058 (0.019) | 0.138 (0.019)

12. Secondary Outcome: Change From Baseline in Pre-BD Forced Expiratory Flow at 25 Percent (%) to 75% (FEF 25-75%) of Forced Vital Capacity (FVC) to Weeks 2, 4, 8, 12, 24, 36, 44, and 52
Description: FEF is the amount of air (in liters) which can be forcibly exhaled from the lungs in the first second of a forced exhalation. FEF 25-75% was defined as the mean FEF between 25% and 75% of the FVC, where FVC was defined as the volume of air (in liters) that can be forcibly blown out after full inspiration in the upright position. Spirometry was performed after a wash out period of bronchodilators according to their action duration.
Time Frame: Baseline (Day 1) to Weeks 2, 4, 8, 12, 24, 36, 44 and 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters/second
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 469 | 466
liters/second
  Week 2 | 0.065 (0.016) | 0.110 (0.016)
  Week 4 | 0.066 (0.015) | 0.115 (0.015)
  Week 8 | 0.069 (0.016) | 0.114 (0.016)
  Week 12 | 0.076 (0.016) | 0.137 (0.016)
  Week 24 | 0.080 (0.017) | 0.142 (0.017)
  Week 36 | 0.087 (0.017) | 0.132 (0.017)
  Week 44 | 0.091 (0.017) | 0.162 (0.017)
  Week 52 | 0.088 (0.017) | 0.135 (0.017)

13. Secondary Outcome: Change From Baseline in Post-BD FEF 25-75% to Weeks 2, 4, 8, 12, 24, 36 and 52
Description: as for outcome 12
Time Frame: Baseline (Day 1) to Weeks 2, 4, 8, 12, 24, 36 and 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters/second
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 469 | 467
liters/second
  Week 2 | 0.074 (0.017) | 0.135 (0.017)
  Week 4 | 0.087 (0.017) | 0.144 (0.017)
  Week 8 | 0.083 (0.017) | 0.144 (0.017)
  Week 12 | 0.089 (0.018) | 0.161 (0.018)
  Week 24 | 0.093 (0.019) | 0.169 (0.019)
  Week 36 | 0.093 (0.019) | 0.161 (0.018)
  Week 52 | 0.093 (0.019) | 0.153 (0.019)

14. Secondary Outcome: Annualized Rate of Severe COPD Exacerbations Over the 52-Week Treatment Period
Description: Moderate exacerbations were recorded by the Investigator and defined as AECOPD that required either systemic corticosteroids (such as intramuscular, intravenous or oral) and/or antibiotics. Severe exacerbations were also recorded by the Investigator and defined as AECOPD requiring hospitalization, or observation for >24 hours in an emergency department/urgent care facility or resulting in death. For both moderate and severe events to be counted as separate events, they were separated by at least 14 days. Annualized event rate was the total number of exacerbations that occurred during the treatment period divided by the total number of participant-years treated. Events were adjudicated by independent third party.
Time Frame: Baseline (Day 1) to Week 52
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: exacerbation per participant-year
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 471 | 468
exacerbation per participant-year | 0.086 [0.050 to 0.147] | 0.072 [0.040 to 0.132]

15. Secondary Outcome: Time to First Moderate or Severe COPD Exacerbation During the 52-Week Treatment Period
Description: The time to first moderate or severe exacerbation was defined as date of the first event minus randomization date +1. The median time to first severe exacerbation was derived from Cox regression model. Moderate exacerbations events were recorded by the investigator and defined as AECOPD that require either systemic corticosteroids (such as intramuscular, intravenous or oral) and/or antibiotics. Severe exacerbations were recorded by the Investigator and defined as AECOPD requiring hospitalization, or observation for >24 hours in an emergency department/urgent care facility or resulting in death. For both moderate and severe events to be counted as separate events, they were separated by at least 14 days.
Time Frame: Baseline (Day 1) and up to Weeks 12, 24, 36 and 52
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 471 | 468
weeks
  Up to Week 12 | 0.019 [0.009 to 0.035] | 0.024 [0.013 to 0.041]
  Up to Week 24 | 0.039 [0.024 to 0.059] | 0.034 [0.021 to 0.054]
  Up to Week 36 | 0.045 [0.029 to 0.067] | 0.039 [0.024 to 0.059]
  Up to Week 52 | 0.061 [0.042 to 0.086] | 0.043 [0.027 to 0.065]

16. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a participant temporally associated with the use of study treatment, whether or not considered related to the study treatment. TEAEs were defined as AEs that developed or worsened in grade or became serious during TE period which was defined as the period from the time of first dose of study treatment until the last visit in the study. Serious adverse events (SAE) were defined as any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event.
Time Frame: TEAEs were collected from the time from the first administration of study treatment to the last administration of the study treatment + 98 days, up to 491 days
Population: The Safety population consisted of all participants who actually received at least 1 dose or partial of a dose of the study treatment, analyzed according to the treatment participants actually received. One participant was exposed to different treatment other than planned (was randomized to placebo arm but received dupilumab on Day 40). The actual arm was considered as dupilumab 300 mg q2w. In safety analyses, the actual arms are used.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 470 | 469
Participants
  Any TEAE | 359 | 365
  Any TESAE | 74 | 65

17. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADA) to Dupilumab
Description: Number of participants with treatment-emergent response to dupilumab with peak post-baseline titers during the on-treatment period are reported. Treatment-emergent response was defined as a positive response in the ADA assay post first dose, when baseline results were negative or missing. Categories were based on titer values and included: low (Titer <1000); moderate (1000<=Titer<=10,000); and high (Titer >10,000). On-treatment period was defined as last study treatment administration plus 14 days; that is, Week 52.
Time Frame: Up to Week 52
Population: The ADA population consisted of all participants in the Safety population with at least 1 reportable ADA results (either 'ADA negative' or 'ADA positive') after first dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 453 | 462
Participants
  Low titer | 7 | 27
  Moderate titer | 0 | 1
  High titer | 0 | 2

ADVERSE EVENTS:
Time Frame: TEAEs were collected from the time from the first administration of study treatment to the last administration of the study treatment + 98 days, up to 491 days
Description: Analysis was performed on the Safety population. One participant was exposed to different treatment other than planned (was randomized to placebo arm but received dupilumab on Day 40). The actual arm was considered as dupilumab 300 mg q2w. In safety analyses, the actual arms are used.
Arm/Group | Placebo | Dupilumab 300 mg q2w
All-Cause Mortality (participants affected / at risk) | 9/470 | 8/469
Serious Adverse Events (participants affected / at risk) | 74/470 | 65/469
Other Adverse Events (participants affected / at risk) | 172/470 | 168/469
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=470) | Dupilumab 300 mg q2w (N=469)
Abdominal Wall Abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Bronchopulmonary Aspergillosis (Infections and infestations) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 4 (4) | 3 (3)
Covid-19 Pneumonia (Infections and infestations) | 5 (5) | 2 (2)
Cholecystitis Infective (Infections and infestations) | 0 (0) | 1 (1)
Epiglottitis (Infections and infestations) | 0 (0) | 1 (1)
Herpes Zoster (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 2 (2) | 3 (4)
Pneumonia (Infections and infestations) | 12 (13) | 6 (7)
Pneumonia Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Pneumococcal (Infections and infestations) | 2 (2) | 0 (0)
Pulmonary Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Septic Shock (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous Abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ductal Adenocarcinoma Of Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung Carcinoma Cell Type Unspecified Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Pancreatic Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous Cell Carcinoma Of Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blood Loss Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaphylactic Reaction (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 1 (2) | 0 (0)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Psychotic Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Basal Ganglia Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral Haemorrhage (Nervous system disorders) | 0 (0) | 2 (2)
Cerebral Infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 1 (2) | 0 (0)
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic Stroke (Nervous system disorders) | 2 (2) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1) | 0 (0)
Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 2 (2) | 1 (1)
Angina Unstable (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular Block Complete (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular Block Second Degree (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Failure (Cardiac disorders) | 2 (2) | 2 (2)
Cardiac Failure Congestive (Cardiac disorders) | 2 (2) | 0 (0)
Cor Pulmonale Acute (Cardiac disorders) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 2 (2)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Nodal Rhythm (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive Crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive Emergency (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Artery Occlusion (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Vascular Disorder (Vascular disorders) | 1 (1) | 0 (0)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 26 (34) | 28 (37)
Chronic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Pneumothorax Spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal Ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal Polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bile Duct Stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic Failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatorenal Syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic Kidney Disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Glomerulonephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Sudden Cardiac Death (General disorders) | 1 (1) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pneumothorax Traumatic (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Rib Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin Abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=470) | Dupilumab 300 mg q2w (N=469)
Nasopharyngitis (Infections and infestations) | 45 (60) | 45 (55)
Upper Respiratory Tract Infection (Infections and infestations) | 46 (66) | 37 (49)
Headache (Nervous system disorders) | 33 (39) | 38 (57)
Hypertension (Vascular disorders) | 28 (32) | 17 (17)
Diarrhoea (Gastrointestinal disorders) | 17 (18) | 25 (34)
Back Pain (Musculoskeletal and connective tissue disorders) | 16 (17) | 25 (27)
Accidental Overdose (Injury, poisoning and procedural complications) | 30 (36) | 26 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-11-07): https://cdn.clinicaltrials.gov/large-docs/32/NCT03930732/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/32/NCT03930732/SAP_001.pdf